CLINICAL TRIAL: NCT03676439
Title: Lateral Cord Magnetic Stimulation For Refractory Spastic Cerebral Palsy - Multicenter Double Blind Randomized and Controlled Trial
Brief Title: Lateral Cord Magnetic Stimulation For Refractory Spastic Cerebral Palsy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sociedad Argenttina de Neuromodulación (Other)
Collaborators: Hospital "San Juan de Dios" - Hurlingham - Argentina (Unknown); Provincial Perogram of Neuromodulation (Pcia Buenos Aires) Argentina (Unknown)
Responsible Party: Principal Investigator, Juan Carlos M. Andreani MD, MD, Sociedad Argenttina de Neuromodulación
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Andreani, JCM 3
Record Dates: First submitted 2018-09-04; First posted 2018-09-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Spastic Cerebral Palsy; Dysarthria
Keywords: Lateral Cord Stimulation; Disability; Magnetic Stimulation; Spasticity; Spinal Cord Stimulation
MeSH Terms: conditions — Cerebral Palsy; Dysarthria; Muscle Spasticity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: A comparision, Randomized and double blinded study
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and independent evaluator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated Arm: Magnetic Spinal Stimulation plus PKT (Active Comparator): Three months of kinesthetic and phoniatric treatment, and Magnetic Spinal Stimulation, 80% of the cervical muscles's motor threshold, 100 pulses at 10Hz, lasting 10 seconds, repeated during 30 minutes, twice a week for 3 months on cervical lateral location, focalized on the Lateral Spinal Cord.
  Interventions: Device: Magnetic Spinal Stimulation
- Sham comparator (Placebo Comparator): They will receive kinesthetic and phoniatric treatment, and during 3 months,with equal periodicity, they will receive a sensible false magnetic stimulation, of equal localization that other arm, with insufficient intensity, to blind clinical experience.
  Interventions: Device: Magnetic Spinal Stimulation

INTERVENTIONS:
Device: Magnetic Spinal Stimulation — Spinal Magnetic Stimulation (TMS) on Lateral Cord Stimulation (LCS), in the search of the improvement of the tone, motor function and speech, in patients with spastic cerebral Palsy.
  Due to its non-invasiveness and possible efficacy, the use of Magnetic Spinal Stimulation is proposed to try to prove its therapeutic usefulness.
  This is the phase 2/3 clinical test of the method, in the future, and as its use could be extended, if the results were positive, its indications could be extended to other pathological conditions, giving a greater spectrum of spastic patients, potentially benefited.
  Other Names: Neuromodulation

SUMMARY:
Lateral cord stimulation (LCS) was discovered by the author as the producer of an average threshold increase for abnormal muscle contraction responses, in experimental pathological conditions, as described and referred.

This physiological effect is proposed to improve tone, motor function and speech, in patients with spasticity of different causes, such as cerebrovascular accident, congenital brain malformations, perinatal anoxia (image called cerebral palsy), sequels of neurosurgery, etc.

Due to its non-invasiveness and possible efficacy, the use of magnetic stimulation is proposed to try to demonstrate its therapeutic utility.

This is the clinical test of phase 2/3 of the method, in the future, and how its use could be extended, if the results were positive, its indications could be extended to other pathological conditions, giving a greater spectrum of spastic patients, potentially benefited

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a chronic and non-progressive morbid disease that affects psychomotor development, with multiple etiologies that share a common condition of acquired perinatal anomalies during development.

The manifestations are multiple and varied, with more frequent motor disorders, speech disorders, mental retardation, spasticity, dystonia, etc.. About a third of these patients have a normal IQ, for whom those signs are more disabling than for others, and for refractory speech problems there is no therapy available These subjects have generally been unsuccessfully treated with medications, botulinum toxin injections, rehabilitation or kinesic orthosis, maintaining their abnormal stable conditions at the end of childhood or early adulthood.

The rational for this clinical trial is that the author has demonstrated the reduction of the excitability threshold of the nociceptive response by electrically stimulating the lateral spinal cord in an animal model, therefore, its possible beneficial action on abnormal muscle tone, somatic motor functions and improvement of speech, by this method.

Spastic Cerebral Palsy has been chosen as a targeted population, because it use to be a chronic and irreversible condition with few therapeutic options, ineffective and frequent complications.

It is of ancient knowledge that electric currents can alter the functions of the Nervous System In the last decades there was a refinement of these techniques of stimulation, being able to emphasize especially the Transcranial or Spinal Magnetic Stimulation (TMS). This therapeutic method, developed in the eighties, is able to modulate brain activity, through the stimulation of limited cortical or spinal areas, with minimal side effects, which is applied through a coil that produces an alternating electrical current.

The constant change of orientation of this alternating current generates a powerful electromagnetic field, capable of crossing the cranial scalp and the skull bone or the osteo-ligamentary structures and originating an electric current restricted to small areas of the brain, cerebellum or spinal cord The objective of the present clinical trial is to demonstrate the therapeutic effect of focal stimulation of the spinal cord in speech and motor function assessed by Modifyied Aschworth sacale and speech, evaluated through Functional Independence Measure (FIM) Scale, selected cases of spastic CP The rational is to focus the magnetic impact on the lateral surface of the spinal cord, trying to stimulate the spinocerebellar tracts, because of its superficial location, therefore, more accessible.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older.
* Spastic Cerebral Palsy with stable condition.
* Motor disability unilateral or predominantly unilateral.
* Clinically evident speech disorders.
* Normal or slightly subnormal intellectual coefficient (I.Q 80 or more)
* Absence of psychiatric disorders

Exclusion Criteria:

* Cardiac or severe respiratory disorders.
* Steady abnormal postures (except possible orthopedic surgical correction)
* Recurrent chronic bronchial or pulmonary infections.
* Psychiatric disorders
* Chronic recurrent urinary infections
* Severe osteoporosis in affected limbs
* Chronic skin ulcers
* Drug addiction.
* Episodes of Status Epileptucus
* Personal history, or in close relatives, of medical legal complaint

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Changes in Modified Ashworth Scale (MAS) | One pre interventional and monthly - up to three months - post interventional
  Scale evaluationg muscle stiffness, from 0(normal) to 5 (maximal rigidity). It wiil be employed to evaluate the spasticity related to limbs.
Changes in Functional Independence measure (FIM) for the speech. | One pre interventional and monthly - up to three months - post interventional
  The FIM measures what an individual can perform - Only the ability for communication, comprehension and expression, will be evaluated to assess speech changes

SECONDARY OUTCOMES:
Changes in Barthel's Scale | One pre interventional and monthly - up to three months - post interventional
  The Barthel Index for Activities of Daily Living (ADL) assesses functional independence, into 10 activities of daily living. Values range from 0 -100, will be investigated to evaluate whole functional changes

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos M Andreani, MD, Study Director — CENIT Foundation & Sociedad Argentina de Neuromodulación; Werner Braunsdorf, MD, Principal Investigator — Klinik von Magdeburg - Germany; Wojciech Maksymowicz, MD, Principal Investigator — University of Warmia and Mazury in Olsztyn- Poland; Tommaso Tufo, MD, Principal Investigator — Policlinico A. Gemelli University Hospital Foundation - Rome - Italy
Locations (1):
- Centro de Rehabilitación San Juan de Dios, Hurlingham, Buenos Aires, Argentina

REFERENCES:
- [Background] Andreani JC, Guma C. Lateral cord stimulation decreases spastic electromyographic spreading: responses in a brain-damaged pig preparation. Neuromodulation. 2008 Jul;11(3):202-7. doi: 10.1111/j.1525-1403.2008.00167.x. PMID 22151097
- [Background] Abdeen MA, Stuchly MA. Modeling of magnetic field stimulation of bent neurons. IEEE Trans Biomed Eng. 1994 Nov;41(11):1092-5. doi: 10.1109/10.335848. PMID 8001998
- [Background] Andreani, JCM, Guma C. Lateral Cord Stimulation (LCS) to relieve spasticity experimental protocol and results. Proceedings of the 10th Conference of the International Federation of Electrical Stimulation (IFESS) Montreal-Canada, July 4-8th 2005. pp 153-5.
- [Background] Duchenne de Boulogne. De l'électrisation localisée et de son application à la physiologie, à la pathologie et à la thérapeutique (3e édition). Librairie JB Bailiere et fils. Paris. 1872.
- [Background] Koy A, Pauls KA, Flossdorf P, Becker J, Schonau E, Maarouf M, Liebig T, Fricke O, Fink GR, Timmermann L. Young adults with dyskinetic cerebral palsy improve subjectively on pallidal stimulation, but not in formal dystonia, gait, speech and swallowing testing. Eur Neurol. 2014;72(5-6):340-8. doi: 10.1159/000360984. Epub 2014 Oct 14. PMID 25322688
- [Background] Lefaucheur JP. Methods of therapeutic cortical stimulation. Neurophysiol Clin. 2009 Feb;39(1):1-14. doi: 10.1016/j.neucli.2008.11.001. Epub 2008 Nov 29. PMID 19268842